

### STATISTICAL REPORTING AND ANALYSIS PLAN

# A RANDOMIZED, 8 WEEK CLINICAL STUDY TO EVALUATE THE EFFICACY OF AN EXPERIMENTAL STANNOUS FLUORIDE DENTIFICE IN THE RELIEF OF DENTINAL HYPERSENSITIVITY

**Protocol Number: 208153** 

Phase: N/A

Property of GSK Consumer Healthcare
Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of GSK
Template Version Effective: 15-Jul-2017
Page 1 of 48

# **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Final Analysis Plan | 14-Dec-2017 | Not applicable (N/A) |

| Та | | f <b>conten</b><br>ment Hist | <b>nts</b><br>tory | 2 |
|---|---|---|---|---|
| | | | nts | |
| 1 | | | ey Protocol Information | |
| | 1.1 | • | Design | |
| | 1.2 | • | Objectives | |
| | 1.3 | • | ent | |
| | 1.4 | | Size Calculation | |
| 2 | Plann | ed Analys | ses | 9 |
| | 2.1 | Interim | Analysis | 9 |
| | 2.2 | Final A | nalyses | 9 |
| 3 | Consi | derations | for Data Analyses and Data Handling Conventions | 10 |
| | 3.1 | Baseline | e Definition | 10 |
| | 3.2 | Subgrou | ups/Stratifications | 10 |
| | 3.3 | Centers | Pools | 10 |
| | 3.4 | Timepo | ints and Visit Windows | 10 |
| 4 | Data Analysis | | | 10 |
| | 4.1 | Populat | ions for Analysis | 11 |
| | | 4.1.1 | Subject Disposition | 11 |
| | | 4.1.2 | Protocol Deviations | 11 |
| | | 4.1.3 | Analysis Populations | 12 |
| | 4.2 | Subject | Demographics and Other Baseline Characteristics | 13 |
| | | 4.2.1 | Demographic Characteristics | 13 |
| | | 4.2.2 | General Medical History | 13 |
| | 4.3 | Study P | roduct Compliance and Use of Other Therapy | 13 |
| | | 4.3.1 | Study Product Compliance and Exposure | 13 |
| | | 4.3.2 | Prior and Concomitant Medication | 13 |
| | | 4.3.3 | Other Therapy/Rescue Medication | 14 |
| | 4.4 | Analysi | s of Efficacy | 14 |
| | | 4.4.1 | Primary Efficacy Endpoint | 14 |
| | | 4.4.2 | Secondary Efficacy Variables | 15 |
| | | 4.4.3 | Handling of Missing Values/Censoring/Discontinuations | 15 |
| | 4.5 | Analysi | s of Secondary Objectives | 15 |
| | | 4.5.1 | Efficacy (Secondary) | 15 |
| | | | Glavo Smith Kline Consumer Healthcare Confidential | |

| | | 4.5.2 | Pharmacokinetic (Secondary) | 16 |
|----|--------|-------------|--------------------------------------------|----|
| | 4.6 | Analysi | is of Exploratory Objectives | 16 |
| | 4.7 | Analysi | is of Safety | 17 |
| | | 4.7.1 | Adverse Events and Serious Adverse Events | 17 |
| | 4.8 | Analysi | is of Other Variables | 18 |
| 5 | Char | nges to the | Protocol Defined Statistical Analysis Plan | 18 |
| | | 5.1.1 | Prior and Concomitant Medication | 19 |
| 6 | Top- | line Sumn | nary | 20 |
| At | tachme | ent 1: List | of Data Displays | 21 |
| | Appe | endix 1: T | emplates for Tables, Figures & Listings | 22 |

# **Abbreviations**

| Abbreviation | Definition |
|-------------------|-------------------------------------|
| AE | Adverse Event |
| ANCOVA | Analysis Of Covariance |
| BDRM | Blinded Data Review Meeting |
| CI | Confidence Interval |
| DH | Dentinal Hypersensitivity |
| eCRF | Electronic Case Report Form |
| GCS | Global Clinical Supplies |
| GSKCH | GlaxoSmithKline Consumer Healthcare |
| ITT | Intent-To-Treat |
| MedDRA | Medical Dictionary For Regulatory |
| N | Number Of Subjects |
| NAF | Sodium Fluoride |
| OST | Oral Soft Tissue |
| PP | Per Protocol |
| ppm | Parts Per Million |
| RLR | Review Listing Requirement |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SE | Standard Error |
| SMFP | Sodium Monofluorophosphate |
| SnCl <sub>2</sub> | Stannous Chloride |
| SnF <sub>2</sub> | Stannous fluoride |
| SOC | System Organ Class |
| w/w | Weight/Weight |

The purpose of this Statistical Reporting and Analysis Plan is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 208153.

## 1 Summary of Key Protocol Information

The purpose of this trial is to demonstrate the efficacy and safety of a experimental 0.454% weight/weight (w/w) Stannous fluoride (SnF<sub>2</sub>) dentifrice to treat the symptoms of Dentinal Hypersensitivity (DH). Efficacy will be demonstrated as a treatment difference in favour of the 0.454% w/w SnF<sub>2</sub> dentifrice versus the Negative Control dentifrice for the primary efficacy outcome, Schiff sensitivity score at Week 8. Safety will be demonstrated through assessment of adverse events (AEs).

#### 1.1 Study Design

#### **Overall Design**

This will be a single centre, randomized, controlled, examiner-blind, 3 treatment arm, parallel group design study, stratified by maximum baseline Schiff sensitivity score (of the 2 selected test teeth), with a treatment period of 8 weeks, to investigate the clinical effectiveness of an experimental SnF<sub>2</sub> dentifrice in the reduction of DH. DH will be assessed at Baseline, and after 4 and 8 weeks treatment.

The study will be conducted in healthy subjects with pre-existing self-reported and clinically diagnosed tooth sensitivity at Screening, in a Chinese population.

An acclimatization period of 2-6 weeks will be included in this study, given that 2 weeks is understood to be an expected amount of time to minimize the potential for carry over effects from prior use of anti-sensitivity products.

In line with Chinese Ministry of Health guidelines [Ministry of Health (China), 2010] for the testing of functional dentifrices (desensitizing), a standard fluoride dentifrice with no specific anti-sensitivity, anti-gingivitis and anti-plaque activity (Chinese marketed Colgate Triple Protection) will be included as the negative control (Negative Control). A Chinese marketed positive control (Positive Control) dentifrice with sensitivity benefits (Crest 7-Effects Strengthen Dental Enamel toothpaste, containing stannous chloride (SnCl<sub>2</sub>)) will also be included in this study design as a benchmark of performance in the Chinese population.

# 1.2 Study Objectives

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| • To compare the clinical efficacy of an experimental 0.454% w/w SnF <sub>2</sub> dentifrice for the relief of DH, as elicited by an evaporative air stimulus (with Schiff sensitivity score), against | • Change from baseline in Schiff sensitivity score at 8 weeks. |

| Objectives | Endpoints |
|---|---|
| a negative control dentifrice, when | |
| used twice daily for 8 weeks. | |
| Secondary Objectives | Secondary Endpoints |
| • To compare the clinical efficacy of an experimental 0.454% w/w SnF <sub>2</sub> dentifrice for the relief of DH, as elicited by a tactile stimulus (Yeaple probe), against a negative control dentifrice, when used twice daily for 8 weeks. | Change from baseline in tactile threshold (Yeaple probe) at 8 weeks. |
| Exploratory Objectives | Exploratory Endpoints |
| • To compare the clinical efficacy of an experimental 0.454% w/w SnF <sub>2</sub> dentifrice for the relief of DH, as elicited by an evaporative air stimulus (with Schiff sensitivity score), against a positive control dentifrice, when used twice daily for 4 and 8 weeks. | Change from baseline in Schiff sensitivity score at 8 weeks. |
| • To compare the clinical efficacy of an experimental 0.454% w/w SnF <sub>2</sub> dentifrice for the relief of DH, as elicited by an evaporative air stimulus (with Schiff sensitivity score), against a negative control dentifrice, when used twice daily for 4 weeks. | Change from baseline in Schiff sensitivity score at 4 weeks. |
| • To compare the clinical efficacy of an experimental 0.454% w/w SnF <sub>2</sub> dentifrice for the relief of DH, as elicited by a tactile stimulus (Yeaple probe), against a negative control dentifrice, when used twice daily for 4 weeks. | Change from baseline in in tactile<br>threshold (Yeaple probe) at 4 weeks. |
| • To compare the clinical efficacy of an experimental 0.454% w/w SnF <sub>2</sub> dentifrice for the relief of DH, as elicited by a tactile stimulus (Yeaple probe), against a positive control dentifrice, when used twice daily for 4 and 8 weeks. | Change from baseline in tactile threshold (Yeaple probe) at 4 and 8weeks. |
| To compare the clinical efficacy of a positive control dentifrice for the relief of DH, as elicited by a tactile | • Change from baseline in tactile threshold (Yeaple probe) at 4 and 8weeks. |

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

| Objectives | Endpoints |
|---|---|
| stimulus (Yeaple probe), against a negative control dentifrice, when used twice daily for 4 and 8 weeks. • To compare the clinical efficacy of a positive control dentifrice for the relief of DH, as elicited by an evaporative air stimulus (with Schiff sensitivity score) against a negative control dentifrice, when used twice daily for 4 and 8 weeks | Change from baseline in Schiff sensitivity score at 4 and 8 weeks. |
| Safety | |
| • To evaluate the safety and oral tolerability of the test dentifrices when used twice daily for 8 weeks. | Adverse Events |

#### 1.3 Treatment

The following study products will be supplied by Global Clinical Supplies (GCS), Glaxosmithkline Consumer Health (GSK CH):

- **Test Product:** Experimental dentifrice containing 0.454% SnF<sub>2</sub> and 0.072% NaF (1450 ppm fluoride in total); CCI
- **Negative Control:** Colgate Triple Protection dentifrice containing 1400 ppm fluoride as sodium monofluorophosphate (SMFP); Chinese Marketplace.
- **Positive Control:** Crest 7-Effects Strengthen Dental Enamel dentifrice containing SnCl<sub>2</sub> and 0.15% NaF (1450 ppm fluoride in total); Chinese marketplace.

Other items to be supplied by the GCS Department, GSK CH:

- **Acclimatization dentifrice:** Colgate Strengthen Fresh Dentifrice containing 1400ppm fluoride as SMFP (Chinese Marketplace).
- Aquafresh Clean Control Toothbrush (UK market place).
- Countdown timers.

#### 1.4 Sample Size Calculation

Change from baseline in Schiff sensitivity score will be used to evaluate treatment effects with regard to the primary objective. With 55 evaluable subjects per group, the study will have 80% power to detect a mean difference of 0.33 (standard deviation [SD]=0.619) in change from baseline in Schiff sensitivity score after 8 weeks of treatment.

The estimate of SD was obtained from GSKCH study 205794. The sample size is based on carrying out 2-tailed 2 sample t-test at a 5% significance level.

Therefore, to allow for dropouts a sufficient amount of subjects will be screened to randomize approximately 180 subjects to ensure 165 subjects (approximately 55 per arm) complete the study.

# 2 Planned Analyses

#### 2.1 Interim Analysis

No interim analysis is planned.

#### 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and database has been locked.

3. All criteria for unblinding the randomization codes have been met and the randomization codes have been distributed

# 3 Considerations for Data Analyses and Data Handling Conventions

#### 3.1 Baseline Definition

For all endpoints, the baseline value will be the latest Day1 (Visit 2) pre-dose assessment with a non-missing value.

Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 3.2 Subgroups/Stratifications

Subgroups are not defined for this trial.

Eligible subjects will be stratified according to their maximum baseline Schiff sensitivity score of the 2 selected teeth. The stratification factor will give rise to 2 strata.

Stratum 1: Maximum Schiff=2. These are subjects with maximum baseline Schiff sensitivity score of 2 for the 2 selected test teeth.

Stratum 2: Maximum Schiff=3. These are subjects with the maximum baseline Schiff sensitivity score of 3 for the 2 selected test teeth.

Efficacy variables will be analyzed accounting for strata.

#### 3.3 Centers Pools

This is a single centre study, therefore pooling of centers is not required.

#### 3.4 Timepoints and Visit Windows

The study schedule should be followed as per protocol. Deviations from the study schedule with respect to visit timings will be reviewed on a case-by-case basis to determine whether the data should be excluded from the Per-Protocol (PP) analysis (Section 4.1.2).

# 4 Data Analysis

Data analysis will be performed by inVentiv Health Clinical. The statistical analysis software used will be SAS version 9.4 (Studio).

Prior to database closure a Blinded Data Review Meeting (BDRM) will be conducted in which various aspects of the trial will be discussed and agreed.

Unless otherwise described below, all listings will be produced for all randomized subjects.

# 4.1 Populations for Analysis

#### 4.1.1 Subject Disposition

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently randomized. A summary will be provided of the number of subjects screened and the number of screen failures with reasons why subjects are not randomized (Table 14.1.1). Percentages for not randomized subjects will be based on number of screened subjects.

Subject disposition will be summarized as the number and percentage of subjects who complete the study, with the number who discontinue broken down by reason for discontinuation (Table 14.1.1). The percentages are based on the total number of subjects randomized. The table will also summarise the number and percent of subjects assigned to each analysis population (defined in Section 4.1.3). The summary will be presented by treatment and overall.

Subject disposition including the subject status (completer, Yes/No), critical demographic data (age, sex, race and ethnicity), the duration of treatment (defined as date of completion or withdrawal minus date of first product application) and the specific reason for discontinuation, will be listed by treatment group for randomized subjects (Listing 16.2.1.1) and non-randomized subjects (Listing 16.2.1.2) separately.

#### 4.1.2 Protocol Deviations

Important major protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed. Details of possible protocol deviation are provided in Protocol Deviation Management Plan (PDMP).

Protocol deviations will be tracked by the study team throughout the conduct of the study. Data will be reviewed prior to unblinding and closure of the database to ensure all important deviations are captured and categorized.

Major deviations of the protocol procedures identified as liable to influence the efficacy outcome may include, but will not be necessarily limited to, the following:

- Violations of inclusion or exclusion criteria that are deemed to affect efficacy
- Medical history which is deemed to affect efficacy.
- Use of prohibited treatment or medication before or during the study, which is felt to affect the assessment of efficacy.
- Not receiving randomised treatment.
- Treatment non-compliance.
- Assessments outside the scheduled time windows.
- Visit outside the planned schedule.
- Protocol deviations.

• Any other reason identified likely to affect efficacy.

Further deviations liable to influence the efficacy outcome will be given in the Review Listing Requirement (RLR) document where major deviations will be identified at the BDRM. The number and percentage of subjects with any major protocol deviation and with each type of major protocol deviations will be presented by treatment (Table 14.1.2) and listed (Listing 16.2.2.1). Any minor protocol deviations will be listed similarly (Listing 16.2.2.2).

#### 4.1.3 Analysis Populations

Five analysis populations are defined.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened<br>Subjects | • All subjects who enter the study and sign the informed consent form. This population includes screen failures as well as those that are randomized. | Disposition, AE listing |
| Randomized | <ul> <li>All subjects who are randomized and may or may not receive dose of the investigational product.</li> <li>Any subject who receives a treatment randomization number will be considered to have been randomized.</li> </ul> | Protocol violations, AE, efficacy, demograp hic characteristic, disposition and medical history listings |
| Safety | <ul> <li>Comprise of all randomized subjects who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | • Safety |
| Intent-To-Treat (ITT) | <ul> <li>Comprise of all randomized subjects who receive at least one dose of study treatment and have at least one post-baseline efficacy evaluation.</li> <li>This population will be based on the treatment to which the subject was randomized.</li> </ul> | • Efficacy |
| Per-Protocol | <ul> <li>All subjects who are assessed as sufficiently compliant with study procedures and restrictions.</li> <li>Subjects with major protocol deviations will be excluded. Depending on the nature of the major protocol deviation and impact on the efficacy variable (s),</li> </ul> | • Efficacy |

| Population | Definition / Criteria | Analyses Evaluated |
|------------|-------------------------------------------|--------------------|
| | subjects will be either completely | |
| | excluded from PP population or only | |
| | partially excluded from the PP analyses. | |
| | This will be determined on a case-by-case | |
| | basis. | |

The primary population for assessment of efficacy will be the ITT Population. A PP analysis will be performed on the primary and secondary efficacy variable if more than 10% of the subjects in the ITT Population are excluded from the PP Population.

Subjects excluded from the analysis populations will be listed (Listing 16.2.3.1).

#### 4.2 Subject Demographics and Other Baseline Characteristics

#### 4.2.1 Demographic Characteristics

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum for continuous variables, and frequency and percentage for categorical variables) will be presented for demographic data by treatment group and overall. These data include age, gender, race, ethnicity and Schiff stratification categories and will be presented for the Safety (Table 14.1.4.1), ITT (Table 14.1.4.2) and if required on the PP Population (Table 14.1.4.3).

Demographic information will be listed (Listing 16.2.4.1) for all randomized subjects.

#### 4.2.2 General Medical History

Medical history data will be listed (Listing 16.2.4.2) with start date and end date or ongoing at the start of study drug. A data listing will also be produced for evaluation of protocol violations at the blinded data review stage.

#### 4.3 Study Product Compliance and Use of Other Therapy

#### 4.3.1 Study Product Compliance and Exposure

Brushing compliance (using study product twice daily) will be presented in the listing (Listing 16.2.5.3) This listing also produced for the blinded data review.

Supervised brushing (subject number, date of visit and time of the supervised procedure and reason why the supervised brushing was not performed according to the protocol) will be listed in the listing (Listing 16.2.5.4). This listings also produced for the blinded data review.

Exposure to the study product will be listed in the listing (Listing 16.1.7)

#### 4.3.2 Prior and Concomitant Medication

Prior treatment will be listed by subject, with, indication, dose, dose form, frequency, route, start date and end date (Listing 16.2.5.1). Prior treatment are defined as those which stopped before the first application of the study product. Concomitant treatment will be listed similarly (Listing 16.2.5.2). Concomitant treatment are defined as those ongoing or started on or after the first application of the study product.

#### 4.3.3 Other Therapy/Rescue Medication

Not Applicable.

### 4.4 Analysis of Efficacy

#### 4.4.1 Primary Efficacy Endpoint

#### 4.4.1.1 Primary Efficacy Endpoint Definition

The change from baseline in Schiff sensitivity score at Week 8 is the primary efficacy endpoint.

The subjects Schiff sensitivity score will be derived as the average score of the 2 test teeth at each visit assessed. The change from baseline will be derived from the individual teeth first before calculating the average change of the 2 test teeth. For post-baseline observations, the average will be calculated only across teeth that have both a valid baseline and a valid post-baseline assessment.

Summary statistics of the observed mean Schiff sensitivity scores and changes from baseline will be presented by treatment at Baseline, Week 4 and Week 8 on the ITT Population (Table 14.2.1.1).

#### 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

The primary analysis is a comparison of the mean change from baseline Schiff sensitivity score between Test Product and Negative Control at Week 8.

The null hypothesis for the primary endpoint is that the mean change from baseline in Schiff sensitivity score is equal between the 2 products.

**H**<sub>0</sub>: 
$$\mu_1 = \mu_2$$

The alternative hypothesis is that the mean change from baseline in Schiff sensitivity score is not equal between the 2 products.

**H**<sub>1</sub>: 
$$\mu_1 \neq \mu_2$$

The change from baseline in Schiff sensitivity score at Week 8 will be analyzed using Analysis of Covariance (ANCOVA) with treatment as factor and mean baseline Schiff sensitivity score as covariate. Note that since the baseline Schiff sensitivity score will be included as a covariate, the baseline Schiff stratification value will not be included in the

GlaxoSmithKline Consumer Healthcare Confidential

model. Adjusted means of all treatments and their standard error (SE), P-value and 95% confidence interval (CIs) will be presented on the ITT Population (Table 14.2.1.2). Treatment differences of the treatment comparisons and SE of it will also be provided together with P-values and 95% CIs.

The assumption of normality and homogeneity of variance in the ANCOVA model will be investigated and if violated, data transformations will be investigated. If suitable transformations cannot be found, non-parametric Van Elteren tests will be performed adjusting for the maximum baseline Schiff sensitivity scores and results will be compared with the ANCOVA results. If the inferences from the 2 analyses are similar then both sets of results will be reported and emphasis will be made on the ANCOVA results. In case of discrepancies between p-values of ANCOVA and Van Elteren analysis, inferences will be drawn on the non-parametric analysis.

To visually inspect the treatment effect on Schiff sensitivity scores, a plot across time (Baseline, Week 4 and Week 8) will be displayed with raw means and SE bars. The plot will display a different symbol line for each treatment group (Figure 14.2.1).

#### 4.4.2 Secondary Efficacy Variables

Secondary efficacy variables are defined in Section 4.5

#### 4.4.3 Handling of Missing Values/Censoring/Discontinuations

Missing data will not be replaced or imputed. Subjects who withdraw from the study prematurely will be included in the statistical analyses up to the point of discontinuation.

#### 4.5 Analysis of Secondary Objectives

#### 4.5.1 Efficacy (Secondary)

#### The change from baseline in tactile threshold at Week 8

The change from baseline in tactile threshold at Week 8 is the secondary efficacy endpoint.

The null hypothesis for the secondary endpoint is that the mean change from baseline in tactile threshold is equal between the 2 products.

H0:  $\mu_1 = \mu_2$ 

The alternative hypothesis is that the mean change from baseline in tactile threshold score is not equal between the 2 products.

H1:  $\mu_1 \neq \mu_2$ 

This secondary efficacy variable analysis will be conducted for the following treatment comparison:

Test Product versus Negative Control at Week 8.

All other treatment comparisons based on the tactile threshold are part of the exploratory objectives.

GlaxoSmithKline Consumer Healthcare Confidential

The subjects tactile threshold will be derived as the average score of the 2 test teeth at each visit assessed and the change from baseline will be derived from the individual teeth first before calculating the average change of the 2 test teeth. If tactile threshold for test teeth is reported as "> 80g" at the post baseline assessments, the value will be taken as as 90g in the derivations.

Summary statistics of the observed mean tactile threshold scores and changes from baseline will be presented by treatment at Baseline, Week 4 and Week 8 (Table 14.2.2.1).

The change from baseline in tactile threshold at Week 8 will be calculated as the subject level mean change from baseline (on the 2 test teeth) and analyzed at Week 8 using ANCOVA with treatment and baseline Schiff stratification value as factors and baseline tactile threshold included as a covariate. Adjusted means of all treatments and their SEs, P-value and 95% CIs will be presented . Treatment differences and SE of all pairs of treatments will be provided together with P-values and 95% CIs (Table 14.2.2.2).

To visually inspect the treatment effect on tactile threshold scores, a plot across time, with the raw means together with SE bars will be produced. The plot will display a different symbol line for each treatment group (Figure 14.2.2).

The assumption of normality and homogeneity of variance in the ANCOVA model will be investigated and if violated, data transformations will be investigated. If suitable transformations cannot be found, non-parametric Van Elteren tests will be performed adjusting for the maximum baseline Schiff sensitivity scores and results will be compared with the ANCOVA results. If the inferences from the 2 analyses are similar then both sets of results will be reported and emphasis will be made on the ANCOVA results. In case of discrepancies between p-values of ANCOVA and van Elteren analysis, inferences will be drawn on the non-parametric analysis.

#### 4.5.2 Pharmacokinetic (Secondary)

Not Applicable

#### 4.6 Analysis of Exploratory Objectives

Exploratory analysis based on the exploratory efficacy variable change from baseline in Schiff sensitivity score and change from baseline in tactile threshold to post baseline (week 4 and 8) will be summarized, analyzed and presented as detailed for the primary and secondary endpoint respectively. Analysis assumptions will be investigated as detailed for the secondary efficacy analysis (Section 4.4.1 and 4.5.1).

The analysis will be conducted for exploratory efficacy variable of Schiff sensitivity scores and tactile threshold for below comparisison (Table 14.2.1.2 and Table 14.2.2.2).

- Test Product versus Negative Control at Week 4
- Test Product versus Positive Control at Week 4 and 8
- Negative Control versus Positive Control at Week 4 and 8

All data for each efficacy variable will be presented for each subject at Baseline, Week 4 and Week 8 (Listing 16.2.6.1 and Listing 16.2.6.2).

#### 4.7 Analysis of Safety

#### 4.7.1 Adverse Events and Serious Adverse Events

All safety data will be reported for the Safety Population as per actual treatment received. The safety profile of the study treatments will be assessed with respect to AEs. Oral soft tissue (OST) abnormalities are included as AEs if they appear or worsen after the initial assessment.

All AEs will be reviewed by the Clinical Research Scientist or Designee prior to database freeze and will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). During this review stage, AEs will be further categorized as oral or non-oral.

AEs will be regarded as treatment-emergent if they occur on or after the first treatment application at the baseline visit.; if this date is missing a suitable alternative will be used eg date of randomization). All other AEs prior to this will be considered non-treatment emergent.

The following summary tables and listings will be presented by treatment group.

- Table of treatment-emergent AEs by system organ class (SOC) and Preferred Term (PT) (Table 14.3.1.1)
- Table of treatment-emergent AEs by Oral/Non-Oral and PT (Table 14.3.1.2)
- Table of treatment-emergent treatment-related AEs by SOC and PT (Table 14.3.1.3)
- Table of treatment-emergent treatment-related serious adverse events (SAEs) by SOC and PT (Table 14.3.1.5) [only produced if there are more than 5 SAEs]
- Table of treatment-emergent treatment-related Non-serious SAEs by SOC and PT (Table 14.3.1.6) [only produced if there are more than 5 SAEs]
- Table of treatment-emergent treatment-related AEs by Oral/Non-Oral and PT (Table 14.3.1.4)
- Listing of all AEs (Listing 16.2.7.1 for all randomized subjects; Listing 16.2.7.2 for non-randomized subjects)
- Listing of deaths (Listing 14.3.2.1)
- Listing of non-fatal SAEs (Listing 14.3.2.2)
- Listing of treatment-emergent AEs leading to study or drug withdrawal (Listing 14.3.2.3)
- Listing of treatment-emergent AEs classified as oral (Listing 14.3.2.4)
- Listing of OST abnormalities (Listing 14.3.2.5)
- Listing of OHT abnormalities (Listing 14.3.2.6)

In the event that there is nothing to report, a null listing will be produced.

#### 4.8 Analysis of Other Variables

To cover the Chinese Ministry of Health guideline requirement, to demonstrate at least a 15% difference between the Test Product and Negative Control, the difference between treatments in the raw means of the actual score (note: not change from baseline) will be calculated using below formula for Schiff sensitivity and tactile threshold at Weeks 4 and 8 (Table 14.2.1.1 and 14.2.2.1).

100\*(Test Product- Negative Control Product)/ Negative Control Product

Similar difference will be calculated between Test product and Positive Control.

### 5 Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in below table

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis section | Statistical Analysis Plan | Rationale for |
| 10.0 ( ) ( ) | 1121 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | Changes |
| <ul> <li>10.2.6. Definition of Analysis Populations • The ITT population includes all randomized subjects who receive at least one dose of investigational product and analysed as randomized. </li> <li>• The PP population includes all subjects who fully comply with all study procedures and restrictions and is a sub-set of the ITT population. Any protocol deviations that would lead to subjects/data being excluded will be removed from the PP</li> </ul> | Comprise of all randomized subjects who receive at least one dose of study treatment and have at least one post-baseline efficacy evaluation. This population will be based on the treatment to which the subject was randomized. All subjects who are assessed as sufficiently compliant with study procedures and restrictions. Subjects with major protocol deviations will be excluded. Depending on the nature of the | To keep consistency across oral studies and to differientate from IIT population definition from safety population. |

| Protocol | | |
|---|---|---|
| Statistical Analysis section | Reporting & Analysis Plan Statistical Analysis Plan | Rationale for Changes |
| population. | major protocol deviation and impact on the efficacy variable (s), subjects will be either completely excluded from PP population or only partially excluded from the PP analyses. This will be determined on a case-by-case basis. | |
| 10.2.1 Demographic and | 4.2.2 General Medical | For medical history |
| <b>Baseline Characteristics</b> | History | and concomitant |
| Descriptive statistics percentages, means and standard deviations) of demographic baseline characteristics, medical history, current/concomitant medication and compliance will be tabulated. | Medical history data will be listed (Listing 16.2.4.2) with start date and end date or ongoing at the start of study drug. 5.1.1 Prior and Concomitant Medication Concomitant medications will be listed by subject, with, indication, dose, dose form, frequency, route, start date and end date | medication coding is not done so listing will be produced. |
| 10.2.5 Safety Analyses | 4.7.1 Adverse Events and | 1) TEAEs by |
| Treatment emergent AEs by SOC, PT and intensity OST abnormalities will be listed and tabulated. The tabulation will show changes in | Serious Adverse Events OST abnormalities will be listed 4.3.1 Study Product Compliance and Exposure | SOC, PT and intensity is study specific and it is decided to not produce for |
| abnormality from baseline to each follow-up assessment. | Exposure to the study product will be listed in the listing | this study 2) In the same listing we |
| Exposure to study product will | | can display |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis section | Statistical Analysis Plan | Rationale for Changes |
| also be tabulated and listed by treatment group. | | the changes in OST 3) To keep consistency across oral studies. |

# **6** Top-line Summary

The outputs required for the topline is summary are documented in the attached worksheet excel file.

# **Attachment 1: List of Data Displays**



# **Appendix 1: Templates for Tables, Figures & Listings**

This is a guideline which will give the guidance of treatment labels that will be used for the table header and in the figures, listings and in the footnotes.

*Note to programmer:* 

- 1) The treatment labels for the column heading will be as follow:
- Test Product
- Negative Control
- Positive Control
- 2) Use following footnotes in all the TLFs:

*Test Product: Dentifrice (0.454% SnF<sub>2</sub> and 0.072% NaF)* 

Negative Control: Dentifrice (1400 ppm F SMFP) Colgate Triple Protection Positive Control: Dentifrice (SnCl<sub>2</sub> and 0.15% NaF 1400 ppm F) Crest 7-Effects

*3) Check actual races captured in eCRF to adjust the race name and abbreviations.* 

Stannous Fluoride (SnF<sub>2</sub>) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

> Table 14.1.1 Subject Disposition All Screened Subjects

Study Population: All Screened Subjects (N=xxx)

| | Test Product<br>(N=XX) | Negative Control<br>(N=XX) | Positive Control<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| TOTAL SUBJECTS SCREENED n (%) | | | | xxx |
| SUBJECTS NOT RANDOMIZED n (%) | | | | Xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | | | | xxx (xx.x) |
| ADVERSE EVENT | | | | Xxx (xx.x) |
| LOST TO FOLLOW UP | | | | xxx (xx.x) |
| PROTOCOL VIOLATION | | | | Xxx (xx.x) |
| WITHDRAWAL OF CONSENT | | | | Xxx (xx.x) |
| OTHER | | | | Xxx (xx.x) |
| UBJECTS RANDOMIZED n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| COMPLETED STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT COMPLETE STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ADVERSE EVENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| LOST TO FOLLOW-UP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WITHDRAWAL OF CONSENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GlaxoSmithKline Consumer Healthcare Confidential

Page 23 of 48

#### Stannous Fluoride (SnF<sub>2</sub>) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

| | Test Product<br>(N=XX) | Negative Control (N=XX) | Positive Control (N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| OTHER | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| SAFETY POPULATION n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ITT POPULATION n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PP POPULATION n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Percentages for non-randomized category are based on number of screened subjects; percentages for randomized category are based on number of randomized subjects

Page x of y

Stannous Fluoride (SnF<sub>2</sub>) 208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Table 14.1.2
Incidence of Major Protocol Deviations
Randomized Population

Study Population: Randomized (N=xxx)

| | Test Product<br>(N=XX) | Negative Control<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| SUBJECTS WITH AT LEAST ONE MAJOR PROTOCOL VIOLATION n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MAJOR PROTOCOL VIOLATIONS NOT<br>LEADING TO EXCLUSION FROM PP<br>n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VIOLATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MAJOR PROTOCOL VIOLATIONS<br>LEADING TO EXCLUSION FROM PP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| n (%)<br>All VISITS | | | | |
| VIOLATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WEEK Y | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VIOLATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Page x of y

Stannous Fluoride (SnF<sub>2</sub>)

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153

# Table 14.1.2.1 Subject Demographics and Baseline Characteristics Safety Population

Program Run Date:xxxx

Study Population: Safety Population (N=XX)

| | Test Product<br>(N=XX) | Negative Control<br>(N=XX) | Positive Control<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| SEX n (%) | | | | |
| MALE | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| FEMALE | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| RACE n (%) | | | | |
| ASIAN | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| BLACK or AFRICAN | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| AMERICAN INDIAN OR ALASKA<br>NATIVE | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| WHITE | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| MULTIPLE | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| ETHNICITY n (%) | | | | |
| HISPANIC OR LATINO | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| NOT HISPANIC OR LATINO | xx (xx.x) | xx (xx.x) | ••• | xx (xx.x) |
| AGE (YEARS) | w. | | | w |
| n | XX | XX<br>- | ••• | XX |

Stannous Fluoride (SnF<sub>2</sub>) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

| | Test Product<br>(N=XX) | Negative Control<br>(N=XX) | Positive Control (N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| MEAN | XX.X | xx.x | ••• | XX.X |
| SD | XX.XX | XX.XX | | xx.xx |
| MEDIAN | XX.X | XX.X | ••• | xx.x |
| MINIMUM | XX | XX | ••• | xx |
| MAXIMUM | XX | XX | ••• | xx |
| STRATIFICATION n (%) | | | | |
| MAXIMUM BASELINE SCHIFF SCORE 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MAXIMUM BASELINE SCHIFF SCORE 3 | | | | |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Page x of y

Stannous Fluoride (SnF<sub>2</sub>) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

# Table 14.2.1.1 Summary Statistics of Evaporative (Air) Schiff Sensitivity Score Intent-to-Treat Population

Study Population: Intent to Treat (N=XXX)

| | | Test P<br>(N= | roduct<br>XX) | | e Control<br>=XX) | Positive Control<br>(N=XX) | | Overall |
|---|---|---|---|---|---|---|---|---|
| Visit | | Observed<br>Value | Change from<br>Baseline | Observed<br>Value | Change from<br>Baseline | Observed<br>Value | Change from<br>Baseline | Observed<br>Value |
| BASELINE | n | XX | | XX | | XX | | XX |
| | n (Missing) | XX | | XX | | XX | | XX |
| | MEAN | x.xx | | X.XX | | x.xx | | X.XX |
| | SE | x.xx | | X.XX | | x.xx | | X.XXX |
| | SD | X.XXX | | X.XXX | | x.xxx | | X.XXX |
| | MEDIAN | x.x | | X.X | | x.x | | X.XX |
| | MINIMUM | x.x | | X.X | | x.x | | X.XX |
| | MAXIMUM | x.x | | X.X | | x.x | | X.X |
| WEEK 4 | n | XX | XX | XX | XX | XX | XX | |
| | n (Missing) | XX | | XX | | XX | | XX |
| | MEAN | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | |
| | SE | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | |
| | SD | X.XXX | x.xxx | X.XXX | x.xxx | x.xxx | X.XXX | |
| | MEDIAN | x.x | x.x | X.X | x.x | x.x | x.x | |
| | MINIMUM | X.X | x.x | X.X | x.x | x.x | x.x | |
| | MAXIMUM | x.x | x.x | X.X | x.x | x.x | x.x | |

Stannous Fluoride (SnF<sub>2</sub>) 208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

| | | Product<br>=XX) | • | e Control<br>=XX) | | Control<br>XX) | Overall |
|---|---|---|---|---|---|---|---|
| Visit | Observed | Change from | Observed | Change from | Observed | Change from | Observed |
| | Value | Baseline | Value | Baseline | Value | Baseline | Value |

WEEK 8 SAME AS WEEK 4.

PPD

Page x of y

Stannous Fluoride (SnF<sub>2</sub>)

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Table 14.2.1.2

Statistical Analysis of Change from Baseline in Evaporative (Air) Schiff Sensitivity Score
Intent-to-Treat Population

Study Population: Intent to Treat (N=XXX)

| | Test Product Negative Control (N=XX) (N=XX) | | Positive Control (N=XX) | |
|---|---|---|---|---|
| WEEK 4 | | | | |
| ADJUSTED MEAN [1] | xx.xx | xx.xx | XX.X | X |
| SE [1] | xx.xxx | XX.XXX | XX.XX | (X |
| 95% CI [1] | (XX.XXX, XX,XXX) | (XX.XXX, XX.XXX) | (XX.XXX, | XX.XXX) |
| P-VALUE [1] | 0.XXXX | 0.XXXX | 0.XXX | X |
| COMPARISONS BETWEEN TREATMENTS | DIFFERENCE (SE) [1] | 95% CI [1] | P-VALUE [1] | MEAN DIFFERENCE % [2] |
| FEST PRODUCT VERSUS NEGATIVE CONTROL [1] * | XX.XX (XX.XXX) | (XX.XXX, XX.XXX) | 0.XXX | xx.xx |
| TEST PRODUCT VERSUS POSITIVE CONTROL [1] | XX.XX (XX.XXX) | (XX.XXX, XX.XXX) | 0.XXX | XX.XX |
| NEGATIVE CONTROL VERSUS POSITIVE CONTROL [1] | XX.XX (XX.XXX) | (XX.XXX, XX.XXX) | 0.XXX | |
| WEEK 8 (AS ABOVE FOR WEEK 4) | | | | |

<sup>\*</sup> Test Product versus Negative Control at Week 8 is a primary endpoint comparision.

Page x of y

<sup>[1]</sup> From ANCOVA model with treatment as factor and baseline Schiff score as covariate. Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment.

<sup>[2]</sup> For the Chinese Ministry of Health guideline requirement to demonstrate difference between Test Product and Control (Positive or Negative) in the observed raw means. It is Calculated as 100\*(Test Product- Control)/Control.

Stannous Fluoride (SnF<sub>2</sub>) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Programming Note: For Table 14.2.2.2 and 14.2.2.4: please update footnote [1] as
[1] From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline tactile threshold as a covariate. Difference is the first named treatment minus second named treatment such that a positive difference favors the first named treatment.

Stannous Fluoride (SnF<sub>2</sub>)

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Table 14.3.1.1
Treatment Emergent Adverse Event by SOC and Preferred Term
Safety Population

| SOC<br>Preferred Term | Test Product<br>(N=XX) | | Negative Control<br>(N=XX) | Positive Control<br>(N=XX) | Overall<br>(N=XX) | |
|---|---|---|---|---|---|---|
| | n (%) | nAE | n (%) nAE | n (%) nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT<br>LEAST ONE AE | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | XX |
| NUMBER OF SUBJECTS WITH NO<br>AE | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | xx |
| SKIN AND SUBCUTANEOUS TISSUE<br>DISORDERS | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | xx |
| ERYTHEMA | xx (xx.x) | XX | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | XX |
| DERMATITIS | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | xx |
| GASTROINTESTINAL SYSTEM | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | xx |
| ABDOMINAL PAIN | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | XX |
| DRY MOUTH | xx (xx.x) | xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | XX |
| VOMITTING | xx (xx.x) | XX | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) | XX |

Etc

Page x of y

n (%) = Number (percent) of subjects nAE = Number of adverse events.

| Stannous | Fluoride | $(SnF_2)$ |
|----------|----------|-----------|
|----------|----------|-----------|

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Listing 16.1.7
Randomization Information
Randomized Population

Study Population: Randomized (N=xx)
Stratum 1: Maximum Schiff score =2

| Subject | Age/Sex/ | Randomization Number | Planned Randomized | Actual Treatment Received | Date of Randomization |
|---|---|---|---|---|---|
| - · · J - · · | 0 , , | | | | |
| Number | Race/Ethinicity[1] | | Treatment | | |

#### PPD

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.

Stannous Fluoride (SnF<sub>2</sub>)

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Listing 16.2.1.1 Subject Disposition Randomized Population

Study Population: Randomized (N=xx)
Treatment Group: Test Product

| | | Screen | Treatment | | Duration of | | | |
|---|---|---|---|---|---|---|---|---|
| | Age/Sex/Race/ | ing | Start Date | Completion/ | Treatment | | Primary Reason for | |
| Subject | Ethinicity [1] | Date | and Time [2] | Withdrawal Date | (Days) [3] | Completed? | Withdrawal | Further Details [4] |

#### PPD

- [1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.
- [2] Date and time of the brushing with allocated treatment date at baseline visit.
- [3] Duration of treatment defined as date of completion or withdrawal minus date of first study product application
- [4] Further details of reasons for withdrawal.

Page x of y

| Stannous Fluoride (SnF <sub>2</sub> ) |
|---------------------------------------|
| 208153 |

Protocol 208153 Program Run Date:xxxx

Listing 16.2.1.2 Subject Disposition Non-Randomized Subjects

Study Population: Non-Randomized (N=xx)

| Subject<br>Number | Age/Sex/Race/<br>Ethinicity [1] | Screening Date | Reason for Screen Failure | Further Details [2] |
|---|---|---|---|---|
| PPD | | | | |

Page x of y

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.
[2] Further details of reasons for screen failure.

| Protoco | 1 208153 | | | Program Run Date:xxx |
|---|---|---|---|---|
| | | | Listing 16.2.2.1<br>for Protocol Deviations<br>Randomized Population | |
| Study Populatio<br>Treatment Group | n: Randomized (N=xx)<br>: XXXXXX | | | |
| Subject | Sex/Age/Race/<br>Ethinicity [1] | Week(s)Excluded<br>from PP Population | Deviation Reason | |
| PPD | | | | |

Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.

Page x of y
| Stannous Fluoride (SnF <sub>2</sub> ) |
|---------------------------------------|
| 208153 |

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Listing 16.2.2.2
Minor Protocol Deviations
Randomized Population

Study Population: Randomized (N=xx)

Treatment Group: Test Product

Subject Age/Sex/Race/ Visit Deviation Sequence Protocol Deviation
Number Ethinicity [1]

## PPD

Page x of y

PPD

Programming Note for Listing 16.2.2.1: Only list those subjects identified in population definition document as being excluded from the PP population.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.

| Stannous Fluoride (<br>208153<br>Final Statistical Rep | $(SnF_2)$ porting and Analysis plan $V1$ | .0 14 Dec 2017 | | | |
|---|---|---|---|---|---|
| Protocol 208153 | | | | | Program Run Date:xxxx |
| | | Exclus | Listing 16.2.3.1<br>ion from Analysis Population<br>Randomized Population | | |
| Study Population: | Randomized (N=xx) | | | | |
| Subject Number | Age/Sex/Race/ Ethinicity [1] | Safety Population | ITT Population | PP Population | |
| PPD | | | | | |
| | | | lack or African American, I = A<br>Ethinicity: H = Hispanic or La | | |

Programming Note for Listing 16.2.3: This listing is based on population definition document.

| 208153<br>Final Statis | | ınd Analysis p | lan V1.0 14 Dec 20 | 17 | | |
|---|---|---|---|---|---|---|
| Protocol 2 | 08153 | | | | | Program Run Date:xxx |
| | | | | Listing 16.2.4<br>Demographic Charact<br>Randomized Popul | eristics | |
| | lation: Randomi<br>Group: Test Pro | | | | | |
| Subject<br>Number | Age (years) | Sex | Race | Ethnicity | Stratum | |
| PPD | | | | | | |

Page x of y

Stannous Fluoride (SnF $_2$ ) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017 Protocol 208153 Listing 16.2.4.2 Medical History and Current Medical Conditions

Program Run Date:xxxx

Study Population: Randomized (N=xx)

Treatment Group: Test Product

Age/Sex/Race/
Subject Ethinicity [1] Any Medical History? Medical Condition Start Date Ongoing? End Date

PPĎ

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.

Randomized Population

Page x of y

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Listing 16.2.5.2

Concomitant Medications and Significant Non-drug Therapies
Randomized Population

Study Population: Randomized (N=xx)
Treatment Group: Test Product

| Subject | Age/Sex/Race/ | Treatment | Sequence | Reason for | Dose Per | Route of | Frequency | Start Date | End Date/Ongoing |
|---|---|---|---|---|---|---|---|---|---|
| Number | Ethinicity [1] | (GSK Drug | Number | Treatment | Adimin. | Admin. | | (Study Day [2]) | |
| | | Synonym) | | | (Unit) | | | | |

### PPD

Page x of y

PPD

Programming note: sort the listing by subject number, treatment start date.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.

[2] Study day relative to the date of randomization.

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date: DDMMYYYY

Listing 16.2.5.3

Brushing Compliance
All Randomized Population

Treatment Group: Test Product 1

| Subject Number | Age/Sex/Race | Period | Expected Number of | Actual Number Brushing | Compliance [4] |
|---|---|---|---|---|---|
| - | Ethinicity [1] | | Brushing [2] | [3] | |

#### PPD

- [1] Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native,A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White White/Caucasian/European Heritage.
- [2] Expected Number of Brushing = 2\*Number of Days between the Two Visits;
- [3] Actual Number of Brushing = Expected Number Missed brushing + Additional Brushing;
- [4] Compliance = Actual Number / Expected Number \*100 (%)

Page x of y

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date: DDMMYYYY

Listing 16.2.5.4

Supervised Brushing Compliance
All Randomized Population

Treatment Group: Test Product 1

| Subject Number | Age/Sex/Race | Visit | Date and Time | Supervised Brushing | Further Details if |
|---|---|---|---|---|---|
| | Ethinicity [1] | | Supervised brushing | Performed (Y/N) | supervised Brushing is |
| | | | started | | not Performed |

## PPD

[1] Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage.

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Listing 16.2.6.1

Individual Efficacy Data for Schiff Sensitivity Score for Two Test Teeth
Randomized Population

Study Population: Randomized (N=xx)
Treatment Group: Test Product 1

| Subject<br>Number | Age/Sex/Race/<br>Ethinicity [1] | Tooth Number<br>(Universal/FDI) | Timepoint | Score | Subject Level<br>Average | Change from<br>Baseline |
|---|---|---|---|---|---|---|
| | LUMINICITY [1] | (Unitversal/TDI) | | | Average | Dasettile |
| PPD | | | | | | |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.

Page x of y

PPD

Programming Note: 1) Subject level average is based raw values for selected 2 test teeth.
2) Please create a similar listsing for tactile

208153

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153

Program Run Date:xxxx

Listing 16.2.7.1 All Adverse Events Randomized Population

Study Population: Randomized (N=xx)
Treatment Group: Test Product 1

| Subject<br>Number | Age/Sex/<br>Race/ | Adverse Event<br>(Preferred Term) | Start Date<br>/Study | Start<br>Time | End<br>Date | End<br>Time | Frequency<br>/Intensity | Related<br>to Study | Action<br>Taken re | Outcome | Serious? | Withdrew? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Ethinici<br>ty [1] | [System Organ<br>Class] | Day[2] | Time | bucc | 11 | [3] | Product? | Study<br>Product | | | [4] |

### PPD

@@ Adverse events with verbatim text ending in this are classified as Oral AEs.

- [1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple; Ethinicity: H = Hispanic or Latino, NH = Not Hispanic or Latino.
- [2] Study day is the day relative to start of treatment, Day 1 being the day of first treatment.
- [3] INT = Intermittent and SGLE = Single.
- [4] Did subject withdraw from study as a result of this adverse event?

### PPD

Programming Note for Listing 16.2.7.2:

- Repeat the same layout for listing 16.2.7.2
- Population should be used 'Non randomized Subjects'
- The fourth column should be only 'Start Date'

Page x of y

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

- Add footnote 'Only SAEs are collected for non randomized subjects'
- Delete the footnote related to study day and adjust the numbers accordingly.

Protocol 207656 Program Run Date: DDMMYYYY

Listing 14.3.2.5
Oral Soft Tissue Abnormalities
All Randomized Population

Treatment Group: Test Product 1

| Subject | Age/Sex/Race/ | Visit | Date and Time of Area | Condition | Changes In OST Details |
|---|---|---|---|---|---|
| Number | Ethinicity [1] | | Assessment | | from Previouse |
| | | | | | Visit (Y/N) |

PPD

Programming Note: For Listing 14.3.2.6 Please remove 'Change in OHT from Previouse Visit' column from this listing.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native,A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage.

Stannous Fluoride (SnF<sub>2</sub>) 208153 Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Protocol 208153 Program Run Date:xxxx

Figure 14.2.1
Evaporative (Air) Schiff Sensitivity Score by Time and Treatment
Intent to Treat Population

Study Population: Intent-to-Treat (N=XX)



Mean and SE plotted are from summary statistics in T 14.2.1.1 Data points have been offset for clarity.

Final Statistical Reporting and Analysis plan V1.0 14 Dec 2017

Note to programmer: (1) Add 'Baseline', 'Week 4' and 'Week 8' to X-axis (2) Use different symbols and line-styles for three treatments (3) For Figures 14.2.3 & 14.2.4 use 'Per Protocol Population' in header.4. Please make sure that Y-axis scale is 0-3 for Schiff score 5) 1) Please make sure that Y-axis scale is 0-80 g for tactile and leble is "Tactile threshold (g)"

Page x of y